CLINICAL TRIAL: NCT06337526
Title: Identifying Factors Associated With Acute Pain Exacerbation in Children With Complex Regional Pain Syndrome (CRPS): A Novel Research Plan
Brief Title: Predicting Pain Exacerbations in Children With Complex Regional Pain Syndrome (CRPS)
Status: Not yet recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Medeloop.ai (Unknown)
Responsible Party: Principal Investigator, Elliot Krane, Professor Emeritus, Dept of Anesthesiology, Stanford University
Other Study IDs: IRB-71503
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Complex Regional Pain Syndromes
Keywords: Child; Pediatrics; Pain; Neuropathic; CRPS
MeSH Terms: conditions — Complex Regional Pain Syndromes; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children & Adolescents with Active CRPS: Subjects between the ages of 10 and 18 years, who have CRPS diagnosed in a pediatric pain center or clinic and whose CRPS is presently active (i.e. unresolved), of either gender, and any ethnicity or racial group.
  For 6 months subjects will wear an Apple Watch, transmitting physiologic and movement data to the investigators, will photograph their meals for AI analysis of content, and log their pain scores and episodes of pain flares, and independently the investigators will collect weather and environmental data in the subject's location. These data will be analyzed by AI to identify chronologic triggers of pain flares.
  Interventions: Device: Apple Watch v8

INTERVENTIONS:
Device: Apple Watch v8 — Apple Watch used for data collection only

SUMMARY:
objectives: identify physiologic, dietary, and environment triggers of severe pain exacerbations in children with CRPS.

DETAILED DESCRIPTION:
Hypothesis(es) and Aims: Investigators hypothesize that spontaneous exacerbations ("flares") of limb pain caused by CRPS have identifiable and predictable precipitants and timing. The aim of this trial is (1) to aggregate large databases of real-time physiological, psychological, subjective pain, environmental and dietary data and analyze these data with artificial intelligence (AI) to identify temporal precipitants to pain exacerbations, and (2) to identify potential strategies to interrupt the progression of acute pain flares based upon what is learned. Early treatment and strategies to interrupt acute pain flares would have a significant effect on quality of life in this patient population while undergoing treatment and resolution of the ongoing condition.

Design: Design of the study: prospective observational study. Subjects: will be recruited from Stanford's pediatric pain clinic and other like centers nation-wide. Subjects will be issued an Apple Watch and the Medeloop app for data collection. Data collection: Medeloop will collect subjects' electronic medical records (existing and prospective) if subjects sign into the hospital's patient portal through Medeloop.

The Apple Watch will transmit physiologic data to Medeloop in real time for a period of 6 months to derive physiologic parameters from Apple Watch measured pulse rate, oxygen saturation, time in daylight, ECG measurement, and movement/activity. Derived variables include heart rate variability, sleep hours, daily distance walked, right/left weight bearing and gait and others. Using a paired smartphone, subjects will photograph all meals for analysis of the dietary content by AI, which will be transmitted to Medeloop after capture for AI analysis. Medeloop software will use location data and cross-reference corresponding environmental and weather data (e.g., atmospheric conditions, air and water quality) on a daily basis. All pain flares will be recorded in real time via the Medeloop app.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of...

Exclusion Criteria:

-

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents with CRPS diagnosed in a pediatric pain management clinic.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pain score | Baseline through month 6
  Pain assessed on an 11-point Likert Scale (score range: 0 to 10)

CONTACTS AND LOCATIONS:
Overall Officials: ANDREW DINH, MD, Principal Investigator — Stanford University; ELLIOT KRANE, MD, Study Director — Stanford University
Locations (1):
- Pediatric Pain Clinic, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abu-Arafeh H, Abu-Arafeh I. Complex regional pain syndrome in children: incidence and clinical characteristics. Arch Dis Child. 2016 Aug;101(8):719-23. doi: 10.1136/archdischild-2015-310233. Epub 2016 Mar 22. PMID 27005945
- [Background] Harden RN, McCabe CS, Goebel A, Massey M, Suvar T, Grieve S, Bruehl S. Complex Regional Pain Syndrome: Practical Diagnostic and Treatment Guidelines, 5th Edition. Pain Med. 2022 Jun 10;23(Suppl 1):S1-S53. doi: 10.1093/pm/pnac046. PMID 35687369
- [Background] Schwartzman RJ, Erwin KL, Alexander GM. The natural history of complex regional pain syndrome. Clin J Pain. 2009 May;25(4):273-80. doi: 10.1097/AJP.0b013e31818ecea5. PMID 19590474
- [Background] Walco GA, Dworkin RH, Krane EJ, LeBel AA, Treede RD. Neuropathic pain in children: Special considerations. Mayo Clin Proc. 2010 Mar;85(3 Suppl):S33-41. doi: 10.4065/mcp.2009.0647. PMID 20194147

DOCUMENTS (1):
  • Informed Consent Form (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT06337526/ICF_000.pdf